CLINICAL TRIAL: NCT06983951
Title: Exploratory Clinical Study Evaluating the Safety and Efficacy of Targeted BCMA Autologous CART Cell Injection in Subjects With Recurrent/Refractory Light Chain Amyloidosis
Brief Title: Exploratory Clinical Study on the Safety and Efficacy of Targeted BCMA Autologous CART Cell Injection in Subjects With Recurrent/Refractory Light Chain Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2024-025
Record Dates: First submitted 2025-02-19; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-02

CONDITIONS: Light Chain Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART (Experimental)
  Interventions: Genetic: BCMA CART

INTERVENTIONS:
Genetic: BCMA CART — The cell product used in this study is a targeted BCMA autologous CART cell injection.
  Research drug name: Targeted BCMA Autologous CART Cell Injection Drug code: BJBR-BCMA-006 Administration method: single intravenous injection

SUMMARY:
This study is a multicenter, open label, fixed dose exploratory clinical trial with an expected enrollment of 30 subjects. The main objective is to evaluate the safety of targeted BCMA autologous CART cell injection in the treatment of recurrent or refractory light chain amyloidosis in subjects, preliminarily verify the effectiveness of targeted BCMA autologous CART cell injection in the treatment of recurrent or refractory light chain amyloidosis in subjects, and explore the pharmacokinetic, pharmacodynamic, and immunogenic characteristics of targeted BCMA autologous CART cell injection after reinfusion.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet all inclusion criteria, and only those who do not meet any exclusion criteria can be enrolled

1. Participants must personally sign the informed consent form approved by the ethics committee in writing before the start of the study;
2. The age of the subject is ≥ 18 years old;
3. Diagnosed with light chain amyloidosis through pathological examination;
4. Subjects with recurrent/refractory light chain amyloidosis who have previously received second-line or higher treatment;
5. dFLC > 50mg/L
6. Expected survival period ≥ 12 weeks;
7. ECOG score ≤ 2 points;
8. Female subjects with fertility should agree to take effective contraceptive measures from the date of signing the informed consent form until 365 days after reinfusion. Effective contraceptive measures are defined as abstinence or using contraceptive methods with an annual failure rate of less than 1% as specified in the plan;
9. Prior to enrollment, participants must have appropriate organ function and meet all of the following test results:

9.1 Absolute neutrophil count ≥ 1.0 × 109/L [allowed to use granulocyte colony-stimulating factor (G-CSF) support]; 9.2 Platelet count ≥ 50 × 109/L; 9.3 Hemoglobin ≥ 8 g/dl; 9.4 Bilirubin value ≤ 1.5 x upper limit of normal (ULN); 9.5 ALT or AST ≤ 2.5 times the upper limit of normal (ULN) (with liver involvement ≤ 5 times the upper limit of normal); 9.6 Mayo 2004 Stage I-IIIa participants; 9.7 Stable coagulation function: INR ≤ 1.5, APTT ≤ 1.2 x upper limit of normal (ULN); Basic blood oxygen saturation is greater than 92% in indoor natural air environment.

Exclusion Criteria:

-

Subjects who meet any of the following criteria will be excluded:

1. Subjects who have received the following previous treatments:

   1.1 Individuals who have received gene therapy prior to enrollment; 1.2 Subjects who received live vaccines within 4 weeks prior to enrollment; 1.3 Received other intervention clinical drug treatments within 12 weeks prior to single collection;
2. Patients with central involvement or complete intestinal obstruction;
3. Patients with moderate to severe pleural and peritoneal effusion who are difficult to control with conventional treatment and require continuous catheterization and drainage;
4. Active malignant tumors within the past 5 years, unless they are curable tumors that have been significantly cured, such as basal or squamous cell carcinoma, cervical or breast carcinoma in situ, etc;
5. Subjects with positive hepatitis B B surface antigen (HBsAg) and abnormal detection of HBV DNA in peripheral blood (abnormal detection of HBV DNA is defined as: quantitative detection of HBV DNA is higher than the detection limit of the testing center or higher than the normal reference value range of the testing center or positive qualitative detection of HBV DNA); Individuals with positive hepatitis C virus (HCV) antibodies and positive hepatitis C virus (HCV) RNA in peripheral blood; Individuals who are HIV antibody positive; Individuals who test positive for Cytomegalovirus (CMV) DNA; Positive RPR results in syphilis testing;
6. There are uncontrollable active infections (excluding CTCAE grade 2 urinary and reproductive system infections and upper respiratory tract infections);
7. Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ III), 24-hour dynamic electrocardiogram showing ventricular arrhythmia and atrioventricular block, positive six minute walk test, interventricular septum and left ventricular posterior wall thickness>1.5cm;
8. Hypertensive subjects who cannot be controlled by drug treatment;
9. Previous treatment toxicity reactions have not improved to baseline or ≤ grade 1 (NCI-CTCAE v5.0 version, except for hair loss and clinically insignificant laboratory test abnormalities);
10. Have undergone major surgery within 2 weeks prior to enrollment, or plan to undergo surgery during the waiting period for reinfusion or within 12 weeks after receiving study treatment (excluding planned local anesthesia surgery);
11. Solid organ transplant recipients;
12. Pregnant or lactating women;
13. Subjects with previous central nervous system disorders (such as cerebral aneurysms, epilepsy, stroke, senile dementia, mental illness, etc.) or consciousness disorders;
14. Other researchers have identified unstable systemic diseases, including but not limited to severe liver, kidney, or metabolic diseases that require drug treatment;
15. Known to have life-threatening allergic reactions, hypersensitivity reactions, or intolerance to cellular preparations or their components;
16. Patients diagnosed by researchers as having bleeding, severe thrombosis, or genetic/acquired bleeding and severe thrombosis (including hemophilia, coagulation dysfunction, thrombocytopenia, splenomegaly, etc.), or patients undergoing thrombolytic or anticoagulant therapy; Researchers believe that there are other situations that are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency Of AES, SAES | 0 day to 24 months after treatment
Dose Limiting Toxicity | 0~28 day after treatment

CONTACTS AND LOCATIONS:
Overall Officials: yajing zhang, MD/PhD, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing Gobroad Brond Hospital, Beijing, Beijing Municipality, China